CLINICAL TRIAL: NCT01969812
Title: Patient Satisfaction and Tolerability With the Evie® Slow-Release Insemination Device: Pilot Study
Brief Title: Tolerability and Satisfaction With Evie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Evie 2013
Record Dates: First submitted 2013-10-22; First posted 2013-10-25 (Estimated); Results first posted 2021-11-17 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-10

CONDITIONS: Infertility
Keywords: Infertility; Intrauterine Insemination; Slow-release Insemination; Evie
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Evie Slow-Release Insemination Device (Experimental): Preliminary studies in Europe have shown increased pregnancy rates using slow-release insemination. Evie slow-release insemination device is a device that is FDA approved. This device has been used in Europe, it has not yet been used at Carolinas Medical Center, by the Women's Institute. The technique for using this device involves loading a pump syringe with the prepared sperm, placing a balloon-secured catheter and syringe in the patient's sounded uterus, and connecting the insemination syringe to the catheter. The slow-release insemination occurs for 4 hours after the insertion of the catheter. The removal procedure, which can be performed by the patient if desired, involves deflating the catheter balloon and removing the catheter.
  Interventions: Device: Evie Slow-release Insemination Device
- Traditional Intrauterine Insemination (Active Comparator): Traditional IUI is one of the treatment modalities for infertility that allows sperm to bypass the cervix and shortens the distance to the fallopian tubes for fertilization. The pregnancy rates for IUI with clomiphene citrate for couples with relatively unexplained infertility have been found to be 7.6% (for women 21-39 years old with up to 3 cycles of IUI with clomiphene).
  Interventions: Other: Traditional Intrauterine Insemination

INTERVENTIONS:
Device: Evie Slow-release Insemination Device
  Arms: Evie Slow-Release Insemination Device
Other: Traditional Intrauterine Insemination
  Arms: Traditional Intrauterine Insemination

SUMMARY:
The purpose of this study is to determine patient satisfaction and tolerability of the Evie® slow-release insemination device for US population. Additionally, to assess cramping with the device and to determine pregnancy rates using the slow insemination device compared to standard IUI.

ELIGIBILITY:
The inclusion criteria:

* Infertile women age ≤39 undergoing first IUI cycle for relatively unexplained infertility
* IRB approval and informed consent signed

Exclusion criteria:

* Women <18 or ≥40 years old
* Women with abnormalities of the uterine cavity
* Women with tubal occlusion
* History of documented pelvic adhesions or endometriosis
* Uncorrected ovulatory dysfunction
* Uncorrected thyroid function
* AMH <1 ng/mL
* <5 million total motile sperm expected for insemination in prior analyses or on the day of sperm preparation for insemination

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Hurst, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Women's Institute at Carolinas Medical Center, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Muharib NS, Abdel Gadir A, Shaw RW. Slow release intrauterine insemination versus the bolus technique in the treatment of women with cervical mucus hostility. Hum Reprod. 1992 Feb;7(2):227-9. doi: 10.1093/oxfordjournals.humrep.a137622. PMID 1577936
- [Background] Reindollar RH, Regan MM, Neumann PJ, Levine BS, Thornton KL, Alper MM, Goldman MB. A randomized clinical trial to evaluate optimal treatment for unexplained infertility: the fast track and standard treatment (FASTT) trial. Fertil Steril. 2010 Aug;94(3):888-99. doi: 10.1016/j.fertnstert.2009.04.022. Epub 2009 Jun 16. PMID 19531445
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Short Form-36. Available at www.sf-36.org. Accessed on September 24, 2013.

RESULTS

PARTICIPANT FLOW:
Groups:
- Evie Slow-Release Insemination Device: Preliminary studies in Europe have shown increased pregnancy rates using slow-release insemination. Evie slow-release insemination device is a device that is FDA approved. This device has been used in Europe, it has not yet been used at Carolinas Medical Center, by the Women's Institute. The technique for using this device involves loading a pump syringe with the prepared sperm, placing a balloon-secured catheter and syringe in the patient's sounded uterus, and connecting the insemination syringe to the catheter. The slow-release insemination occurs for 4 hours after the insertion of the catheter. The removal procedure, which can be performed by the patient if desired, involves deflating the catheter balloon and removing the catheter.
  Evie Slow-release Insemination Device
- Traditional Intrauterine Insemination: Traditional IUI is one of the treatment modalities for infertility that allows sperm to bypass the cervix and shortens the distance to the fallopian tubes for fertilization. The pregnancy rates for IUI with clomiphene citrate for couples with relatively unexplained infertility have been found to be 7.6% (for women 21-39 years old with up to 3 cycles of IUI with clomiphene).
  Traditional Intrauterine Insemination
Period: Overall Study
Arm/Group | Evie Slow-Release Insemination Device | Traditional Intrauterine Insemination
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Evie Slow-Release Insemination Device | Traditional Intrauterine Insemination | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 10 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Patient Tolerability and Satisfaction SF36
Description: The primary outcome variable will be patient tolerability and satisfaction, based on a standardized SF-36 survey.
  Total score 0-100 with higher score denoting better outcomes
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Evie Slow-Release Insemination Device | Traditional Intrauterine Insemination
Number analyzed (Participants) | 12 | 10
units on a scale | 76.8 (15.90) | 84.2 (11.28)

2. Secondary Outcome: Cramping
Description: Cramping assessment based on a Numerical Rating Scale 0 to 10. Higher score denotes worse cramping.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Evie Slow-Release Insemination Device | Traditional Intrauterine Insemination
Number analyzed (Participants) | 12 | 10
score on a scale | 3.85 (2.00) | 2.42 (1.93)

3. Secondary Outcome: Pregnancy Rates
Description: Pregnancy rates based on blood and urine beta-HCG.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Evie Slow-Release Insemination Device | Traditional Intrauterine Insemination
Number analyzed (Participants) | 12 | 10
Participants | 4 | 3

ADVERSE EVENTS:
Arm/Group | Evie Slow-Release Insemination Device | Traditional Intrauterine Insemination
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes